CLINICAL TRIAL: NCT01939743
Title: Diclofenac Suppository As a Preemptive Analgesia in Ultrasound Guided Biopsy of Prostate: Randomized Controlled Trial
Brief Title: Efficacy of Diclofenac Suppository for Pain Control in Ultrasound Guided Biopsy of Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Naveed Haroon, Resident, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11GS009SUR
Record Dates: First submitted 2013-04-01; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Carcinoma Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diclofenac suppository plus lidocaine gel (Experimental): Intervention Drug with local anaesthetic
  Interventions: Drug: Diclofenac suppository plus lidocaine gel; Drug: Lidocaine gel only
- Lidocaine gel only (Other): Used as local aneaethetic as a part of institutional prostate biopsy protocol
  Interventions: Drug: Lidocaine gel only

INTERVENTIONS:
Drug: Diclofenac suppository plus lidocaine gel
  Other Names: Voltral suppository
  Arms: diclofenac suppository plus lidocaine gel
Drug: Lidocaine gel only

SUMMARY:
Transrectal ultrasound guided biopsy of prostate (TRUS-Bx) is widely used as accepted mode of investigation for prostate cancer in current urology practice. It is considered a minor procedure, which most of the patients tolerate, however 20% of patients refuse to undergo the redo procedure without any analgesia or anesthesia but on the other hand, some authors reveal that 65 to 90% of patients report pain ranging from mild to severe in intensity. Diclofenac is a local and systemic anti-inflammatory drug and it reduces local mediators involved in local pain.The purpose of this study is to find out the role of rectal administration of diclofenac suppositories as an adjunct to 2% xylocaine gel in alleviating intra and post procedural pain in prostatic biopsy with adequately calculated sample size and excluding the patients with contraindication to procedure or diclofenac administration as these were the shortcomings of previous studies.

ELIGIBILITY:
Inclusion Criteria:All male patients undergoing ultrasound guided prostate biopsy due to any one of the following:

* Raised prostate-specific antigen level (>4.0ng/ml) and palpable nodularity on digital rectal examination
* Palpable nodularity on digital rectal examination
* Hypo echoic lesion as compared to surrounding prostate on transrectal ultrasound

Exclusion Criteria:

* History of previous prostate biopsy
* Acute and/or chronic prostatitis or chronic pelvic pain syndrome
* Anal fissure, hemorrhoids, anal surgery
* Concomitant analgesic medication
* Chronic renal failure
* Allergy to diclofenac

Ages: 51 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pain on visual analog score | Two hours

SECONDARY OUTCOMES:
Adverse effects of diclofenac suppository | two hours

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Haroon, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Irer B, Gulcu A, Aslan G, Goktay Y, Celebi I. Diclofenac suppository administration in conjunction with lidocaine gel during transrectal ultrasound-guided prostate biopsy: prospective, randomized, placebo-controlled study. Urology. 2005 Oct;66(4):799-802. doi: 10.1016/j.urology.2005.04.053. PMID 16230141
- [Background] Haq A, Patel HR, Habib MR, Donaldson PJ, Parry JR. Diclofenac suppository analgesia for transrectal ultrasound guided biopsies of the prostate: a double-blind, randomized controlled trial. J Urol. 2004 Apr;171(4):1489-91. doi: 10.1097/01.ju.0000115706.19605.e4. PMID 15017205